CLINICAL TRIAL: NCT02398786
Title: Myotonic Dystrophy Family Registry
Acronym: MDFR
Status: Recruiting | Type: Observational
Sponsor: Myotonic Dystrophy Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MDF001
Record Dates: First submitted 2015-03-06; First posted 2015-03-26 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Myotonic Dystrophy; Congenital Myotonic Dystrophy; Myotonic Dystrophy 1; Myotonic Dystrophy 2; Dystrophia Myotonica; Dystrophia Myotonica 1; Dystrophia Myotonica 2; Myotonia Dystrophica; Myotonic Dystrophy, Congenital; Myotonic Myopathy, Proximal; PROMM (Proximal Myotonic Myopathy); Proximal Myotonic Myopathy; Steinert Disease; Steinert Myotonic Dystrophy; Steinert's Disease; Myotonia Atrophica
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Patient-entered data — This registry provides patient-entered data for future clinical trial and study use.

SUMMARY:
The Myotonic Dystrophy Family Registry (MDFR) is an online, patient-entered database that collects information on myotonic dystrophy (DM) to aid researchers in developing new, effective treatments and help identify participants for research studies and clinical trials.

DETAILED DESCRIPTION:
The Myotonic Dystrophy Family Registry (MDFR) is an online, patient-entered database that collects information on myotonic dystrophy (DM) such as disease symptoms and demographic information to aid researchers in developing new, effective treatments and help identify participants for research studies and clinical trials.

The Registry supports trials and studies, making it easier for researchers to explore data and identify possible trial and study participants. It is the first DM registry that gives community members the opportunity to explore anonymous Registry data, to see what the DM community looks like and what others with DM experience. It also provides information on the community of people living with DM, giving researchers and other medical professionals the opportunity to improve how they treat those affected with DM and learn more about how and why certain treatments work and don't work.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with congenital, juvenile-onset or adult onset DM1 or DM2 (confirmed by clinical exam or genetic test)

Exclusion Criteria:

* Not diagnosed with DM, unaffected family members

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will volunteer to participate in this study and enter their own information. The study will be advertised through neuromuscular disease clinics and the Myotonic Dystrophy Foundation and Myotonic Dystrophy Family Registry websites.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2013-02; Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcomes | 36 months
  Number of patients reporting specific symptoms and symptom severity, as well as impacts to quality of life and overall burden of disease in order to inform clinical trial development, understanding of disease for academic, industry and federal agency stakeholders and overall policy decisions. Results will be analyzed in comparison to other registry data and surveys to characterize this disease population cohort and to further define the population.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Stevenson, EdD, MPH, Study Chair — Myotonic Dystrophy Foundation
Locations (1):
- Myotonic Dystrophy Foundation, Oakland, California, United States

REFERENCES:
- See also: Myotonic Dystrophy Family Registry (MDFR) Web portal. — https://myotonicregistry.patientcrossroads.org/